CLINICAL TRIAL: NCT02421913
Title: Efficacy of S(+)-Ketamine Administered as a Continuous Infusion for the Control of Postoperative Pain: a Randomized Controlled Trial
Brief Title: Efficacy of S(+)-Ketamine Administered as a Continuous Infusion for the Control of Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Medico Campinas (Other)
Responsible Party: Principal Investigator, LUIZ EDUARDO DE PAULA GOMES MIZIARA, Physician, Centro Medico Campinas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMCampinas
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S(+)-ketamine group (SG) (Active Comparator): Five minutes before surgery, patients in the SG group received an intravenous continuous infusion containing 0.3 mg.kg-1.h-1 of S(+)-ketamine
  Interventions: Drug: S(+)-Ketamine
- placebo group (PG) (Placebo Comparator): PG received the same dose of saline.

INTERVENTIONS:
Drug: S(+)-Ketamine — S(+)-Ketamine 0,3mg/kg/hr intraoperative
  Arms: S(+)-ketamine group (SG)

SUMMARY:
Background: The use of low-dose continuous infusion of S(+)-ketamine combined with target-controlled intravenous anesthesia with remifentanil and propofol may be related to the control of postoperative pain and of opioid-induced hyperalgesia. The present study aimed to evaluate the efficacy of continuous infusion of S(+)-ketamine given intraoperatively in the control of postoperative pain compared to placebo.

DETAILED DESCRIPTION:
Methods: This is a double-blind randomized controlled trial with 48 patients of both genders aged from 18 to 65 years who underwent videolaparoscopic cholecystectomy. After venipuncture, patients received intravenous parecoxib sodium (40 mg). Target-controlled intravenous anesthesia was induced with propofol and remifentanil associated with rocuronium and adjusted to maintain the bispectral index between 35 and 50. The S(+)-ketamine group (SG) group received a continuous infusion of S(+)-ketamine at a dose of 0.3mg.kg-1.h-1, while the placebo group (PG) received a continuous infusion of saline at the same dose. Postoperative analgesia was measured by a verbal numerical scale (VNS) from 0 to 10 during 12 hours and treated with morphine when VNS score was equal to or higher than 3 at a dose of 0.05 mg.kg-1 when the patient reported pain for the first time and at a dose of 0.025mg.kg-1 on subsequent occasions. Pain scores were recorded in the postoperative care unit (PACU) and at 4 and 12 hours after the end of the surgery The amount of morphine used during PACU stay, from PACU discharge to 4 hours after surgery, and from 4 to 12 hours after surgery, the overall dose of morphine used, and possible adverse effects were also assessed

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 65 Years ASA I and II Accepts healthy volunteers.

Exclusion Criteria:

alcohol or illicit drugs, H2 inhibitors, opioids, or calcium-channel blockers within the last 10 days chronic pain, myocardial ischemia, psychiatric diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467
- [Background] Untergehrer G, Jordan D, Eyl S, Schneider G. Effects of propofol, sevoflurane, remifentanil, and (S)-ketamine in subanesthetic concentrations on visceral and somatosensory pain-evoked potentials. Anesthesiology. 2013 Feb;118(2):308-17. doi: 10.1097/ALN.0b013e318279fb21. PMID 23254146
- [Derived] Miziara LE, Simoni RF, Esteves LO, Cangiani LH, Grillo-Filho GF, Paula AG. Efficacy of Continuous S(+)-Ketamine Infusion for Postoperative Pain Control: A Randomized Placebo-Controlled Trial. Anesthesiol Res Pract. 2016;2016:6918327. doi: 10.1155/2016/6918327. Epub 2016 Feb 2. PMID 26949390